CLINICAL TRIAL: NCT00810979
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Safety and Efficacy of Different Doses of SLx-4090 in Combination With a Statin vs. Statin Mono-therapy in Patients With Hyperlipidemia
Brief Title: Comparison of SLx-4090 Combined With Statin Therapy Versus Statin Alone in Reducing LDL-C in Patients With Hyperlipidemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Response Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLx-4090-08-06
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-04

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias | interventions — 6-(4'-trifluoromethyl-6-methoxybiphenyl-2-ylcarboxamido)-1,2,3,4-tetrahydroisoquinoline-2-carboxylic acid phenyl ester; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): SLx-4090 dose #1 in combination with statin drug. Subjects were dosed with the statin prescribed specifically by their prescribing physician.
  Interventions: Drug: SLx-4090; Drug: Statin
- 2 (Experimental): SLx-4090 dose #2 in combination with statin drug. Subjects were dosed with the statin prescribed specifically by their prescribing physician.
  Interventions: Drug: SLx-4090; Drug: Statin
- 3 (Other): Placebo in combination with statin drug. Subjects were dosed with the statin prescribed specifically by their prescribing physician.
  Interventions: Other: Placebo; Drug: Statin

INTERVENTIONS:
Drug: SLx-4090 — tablet
  Arms: 1
Drug: SLx-4090 — tablet
  Arms: 2
Other: Placebo — matching tablet
  Arms: 3
Drug: Statin — Subjects were dosed with the statin prescribed specifically by their prescribing physician.

SUMMARY:
The purpose of this study is to determine whether SLx-4090 in combination with statin therapy will reduce LDL-C in patients with hyperlipidemia more effectively than statin therapy alone.

DETAILED DESCRIPTION:
1. LDL-C after 12 weeks of treatment
2. Safety and tolerability
3. Plasma levels of SLx-4090

ELIGIBILITY:
Inclusion Criteria:

* LDL-C > or = 100 mg/dL
* On stable statin therapy for at least 6 weeks

Exclusion Criteria:

* Coronary heart disease or risk factors for CHD

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Reduction in LDL-C | 12 weeks

SECONDARY OUTCOMES:
Adverse events | 12 weeks

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Birmingham, Alabama
  - Tempe, Arizona
  - Tucson, Arizona
  - Jacksonville, Florida
  - Atlanta, Georgia
  - Addison, Illinois
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - Edina, Minnesota
  - St Louis, Missouri
  - Rochester, New York
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Mt. Pleasant, South Carolina
  - Richmond, Virginia